CLINICAL TRIAL: NCT06364566
Title: Exploring the Optimal Timing of Minimally Invasive Surgery for Esophageal Squamous Cell Carcinoma After Neoadjuvant Chemoradiotherapy
Brief Title: Exploring the Optimal Timing of Minimally Invasive Surgery for Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: time-exploring
Record Dates: First submitted 2024-04-05; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Time

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short interval group (Experimental): The patient underwent minimally invasive esophagectomy within 50 days after receiving neoadjuvant therapy
  Interventions: Radiation: Neoadjuvant chemradiotherapy; Procedure: Minimally invasive esophagectomy
- Long interval group (Experimental): The patient underwent minimally invasive esophagectomy 50 days after receiving neoadjuvant therapy
  Interventions: Radiation: Neoadjuvant chemradiotherapy; Procedure: Minimally invasive esophagectomy

INTERVENTIONS:
Radiation: Neoadjuvant chemradiotherapy — Patients receiving neoadjuvant chemradiotherapy cause tumor shrinkage
Procedure: Minimally invasive esophagectomy — The patient underwent minimally invasive esophagectomy to remove residual tumors and surrounding lymph nodes

SUMMARY:
The optimal interval between neoadjuvant chemradiotherapy and esophagectomy is still a question that needs to be explored for patients with esophageal squamous cell carcinoma. In this study, based on previous studies, the investigators divided patients into two groups with a cutoff value of 50 days. By comparing the overall survival and disease-free survival of the entire population and non PCR population, the investigators ultimately obtained the optimal surgical timing suitable for clinical use

DETAILED DESCRIPTION:
background：Neoadjuvant chemoradiotherapy has gradually become a first-line treatment for esophageal squamous cell carcinoma patients. After the completion of neoadjuvant chemoradiotherapy, patients usually undergo minimally invasive surgery to ensure complete removal of the tumor and lymphatic tissue. However, the optimal interval between neoadjuvant chemoradiotherapy and minimally invasive surgery is still an unknown factor, and whether it affects postoperative disease-free survival (DFS) and overall survival (OS) of patients remains unknown. Therefore, the main purpose of this study is to explore the specific impact of the interval between neoadjuvant chemoradiotherapy and minimally invasive surgery on patients, and to find the optimal interval time.

methods：Patients who underwent neoadjuvant chemoradiotherapy and minimally invasive surgery from two institutions between October 2010 and September 2019 were included in this study. The time interval is defined as the days between the last time a patient receives neoadjuvant chemoradiotherapy and the execution of surgery. Based on past research, the interval between the two groups was determined to be 50 days. The main research result is the OS and DFS of different interval groups in the overall population and non-PCR population. A multivariate Cox regression model was established to determine the main factors affecting Patient's OS and DFS.

ELIGIBILITY:
Inclusion Criteria:

* (I) thoracic ESCC
* (II) no history of concomitant or prior malignancy
* (III) Completed one cycle of nCRT
* (IV) Received endoscopic radical surgery for esophageal cancer

Exclusion Criteria:

* (I)other histological subtypes
* (II)Received ESD treatment
* (III) Radiation dose greater than 50Gy
* (IV) Metastatic esophageal squamous cell carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2010-10-15 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
The overall survival of the overall population | 5 years
  Does the overall population survive
The Disease-Free survival of the overall population | 5 years
  Is there any tumor metastasis or recurrence in the overall population
The overall survival of the non-PCR population | 5 years
  Does the non-PCR population survive
The Disease-Free survival of the non-PCR population | 5 years
  Is there any tumor metastasis or recurrence in the non-PCR population
The overall survival of the PCR population | 5 years
  Does the PCR population survive
The Disease-Free survival of the PCR population | 5 years
  Is there any tumor metastasis or recurrence in the PCR population

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Ohashi S, Miyamoto S, Kikuchi O, Goto T, Amanuma Y, Muto M. Recent Advances From Basic and Clinical Studies of Esophageal Squamous Cell Carcinoma. Gastroenterology. 2015 Dec;149(7):1700-15. doi: 10.1053/j.gastro.2015.08.054. Epub 2015 Sep 12. PMID 26376349
- [Result] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Result] Eyck BM, van Lanschot JJB, Hulshof MCCM, van der Wilk BJ, Shapiro J, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch OR, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Spillenaar Bilgen EJ, van der Sangen MJC, Rozema T, Ten Kate FJW, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS Study Group. Ten-Year Outcome of Neoadjuvant Chemoradiotherapy Plus Surgery for Esophageal Cancer: The Randomized Controlled CROSS Trial. J Clin Oncol. 2021 Jun 20;39(18):1995-2004. doi: 10.1200/JCO.20.03614. Epub 2021 Apr 23. PMID 33891478
- [Result] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Result] Piessen G, Messager M, Mirabel X, Briez N, Robb WB, Adenis A, Mariette C. Is there a role for surgery for patients with a complete clinical response after chemoradiation for esophageal cancer? An intention-to-treat case-control study. Ann Surg. 2013 Nov;258(5):793-9; discussion 799-800. doi: 10.1097/SLA.0000000000000228. PMID 24096755
- [Result] Eyck BM, van der Wilk BJ, Noordman BJ, Wijnhoven BPL, Lagarde SM, Hartgrink HH, Coene PPLO, Dekker JWT, Doukas M, van der Gaast A, Heisterkamp J, Kouwenhoven EA, Nieuwenhuijzen GAP, Pierie JEN, Rosman C, van Sandick JW, van der Sangen MJC, Sosef MN, van der Zaag ES, Spaander MCW, Valkema R, Lingsma HF, Steyerberg EW, van Lanschot JJB; SANO-study group. Updated protocol of the SANO trial: a stepped-wedge cluster randomised trial comparing surgery with active surveillance after neoadjuvant chemoradiotherapy for oesophageal cancer. Trials. 2021 May 17;22(1):345. doi: 10.1186/s13063-021-05274-w. PMID 34001287
- [Result] Petrelli F, Sgroi G, Sarti E, Barni S. Increasing the Interval Between Neoadjuvant Chemoradiotherapy and Surgery in Rectal Cancer: A Meta-analysis of Published Studies. Ann Surg. 2016 Mar;263(3):458-64. doi: 10.1097/SLA.0000000000000368. PMID 24263329
- [Result] Rombouts AJM, Hugen N, Elferink MAG, Nagtegaal ID, de Wilt JHW. Treatment Interval between Neoadjuvant Chemoradiotherapy and Surgery in Rectal Cancer Patients: A Population-Based Study. Ann Surg Oncol. 2016 Oct;23(11):3593-3601. doi: 10.1245/s10434-016-5294-0. Epub 2016 Jun 1. PMID 27251135
- [Result] Verweij ME, Franzen J, van Grevenstein WMU, Verkooijen HM, Intven MPW. Timing of rectal cancer surgery after short-course radiotherapy: national database study. Br J Surg. 2023 Jun 12;110(7):839-845. doi: 10.1093/bjs/znad113. PMID 37172197
- [Result] Delanian S, Lefaix JL. Current management for late normal tissue injury: radiation-induced fibrosis and necrosis. Semin Radiat Oncol. 2007 Apr;17(2):99-107. doi: 10.1016/j.semradonc.2006.11.006. PMID 17395040
- [Result] Chiu CH, Chao YK, Chang HK, Tseng CK, Chan SC, Liu YH, Chen WH. Interval between neoadjuvant chemoradiotherapy and surgery for esophageal squamous cell carcinoma: does delayed surgery impact outcome? Ann Surg Oncol. 2013 Dec;20(13):4245-51. doi: 10.1245/s10434-013-3139-7. PMID 23959050
- [Result] Shapiro J, van Hagen P, Lingsma HF, Wijnhoven BP, Biermann K, ten Kate FJ, Steyerberg EW, van der Gaast A, van Lanschot JJ; CROSS Study Group. Prolonged time to surgery after neoadjuvant chemoradiotherapy increases histopathological response without affecting survival in patients with esophageal or junctional cancer. Ann Surg. 2014 Nov;260(5):807-13; discussion 813-4. doi: 10.1097/SLA.0000000000000966. PMID 25379852
- [Result] Nilsson K, Klevebro F, Rouvelas I, Lindblad M, Szabo E, Halldestam I, Smedh U, Wallner B, Johansson J, Johnsen G, Aahlin EK, Johannessen HO, Hjortland GO, Bartella I, Schroder W, Bruns C, Nilsson M. Surgical Morbidity and Mortality From the Multicenter Randomized Controlled NeoRes II Trial: Standard Versus Prolonged Time to Surgery After Neoadjuvant Chemoradiotherapy for Esophageal Cancer. Ann Surg. 2020 Nov;272(5):684-689. doi: 10.1097/SLA.0000000000004340. PMID 32833767
- [Result] van der Wilk BJ, Noordman BJ, Neijenhuis LKA, Nieboer D, Nieuwenhuijzen GAP, Sosef MN, van Berge Henegouwen MI, Lagarde SM, Spaander MCW, Valkema R, Biermann K, Wijnhoven BPL, van der Gaast A, van Lanschot JJB, Doukas M, Nikkessen S, Luyer M, Schoon EJ, Roef MJ, van Lijnschoten I, Oostenbrug LE, Riedl RG, Gisbertz SS, Krishnadath KK, Bennink RJ, Meijer SL; Collaborators:. Active Surveillance Versus Immediate Surgery in Clinically Complete Responders After Neoadjuvant Chemoradiotherapy for Esophageal Cancer: A Multicenter Propensity Matched Study. Ann Surg. 2021 Dec 1;274(6):1009-1016. doi: 10.1097/SLA.0000000000003636. PMID 31592898
- [Result] Chidambaram S, Owen R, Sgromo B, Chmura M, Kisiel A, Evans R, Griffiths EA, Castoro C, Gronnier C, MaoAwyes MA, Gutschow CA, Piessen G, Degisors S, Alvieri R, Feldman H, Capovilla G, Grimminger PP, Han S, Low DE, Moore J, Gossage J, Voeten D, Gisbertz SS, Ruurda J, van Hillegersberg R, D'Journo XB, Chmelo J, Phillips AW, Rosati R, Hanna GB, Maynard N, Hofstetter W, Ferri L, Berge Henegouwen MI, Markar SR. Delayed Surgical Intervention After Chemoradiotherapy in Esophageal Cancer: (DICE) Study. Ann Surg. 2023 Nov 1;278(5):701-708. doi: 10.1097/SLA.0000000000006028. Epub 2023 Jul 21. PMID 37477039
- [Result] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Result] Yun JK, Chong BK, Kim HJ, Lee IS, Gong CS, Kim BS, Lee GD, Choi S, Kim HR, Kim DK, Park SI, Kim YH. Comparative outcomes of robot-assisted minimally invasive versus open esophagectomy in patients with esophageal squamous cell carcinoma: a propensity score-weighted analysis. Dis Esophagus. 2020 May 15;33(5):doz071. doi: 10.1093/dote/doz071. PMID 31665266
- [Result] Klevebro F, Nilsson K, Lindblad M, Ekman S, Johansson J, Lundell L, Ndegwa N, Hedberg J, Nilsson M. Association between time interval from neoadjuvant chemoradiotherapy to surgery and complete histological tumor response in esophageal and gastroesophageal junction cancer: a national cohort study. Dis Esophagus. 2020 May 15;33(5):doz078. doi: 10.1093/dote/doz078. PMID 31676895
- [Result] Gakuhara A, Yamashita K, Miyazaki Y, Adachi K, Momose K, Saito T, Tanaka K, Makino T, Yamamoto K, Takahashi T, Kurokawa Y, Nakajima K, Eguchi H, Doki Y. Association between fibrosis around the tumor and postoperative infectious complication in patients with esophageal cancer who underwent preoperative therapy. World J Surg. 2024 Apr;48(4):914-923. doi: 10.1002/wjs.12100. Epub 2024 Feb 6. PMID 38319155
- [Result] Kim JY, Correa AM, Vaporciyan AA, Roth JA, Mehran RJ, Walsh GL, Rice DC, Ajani JA, Maru DM, Bhutani MS, Welsh J, Marom EM, Swisher SG, Hofstetter WL. Does the timing of esophagectomy after chemoradiation affect outcome? Ann Thorac Surg. 2012 Jan;93(1):207-12; discussion 212-3. doi: 10.1016/j.athoracsur.2011.05.021. Epub 2011 Oct 1. PMID 21962263
- [Result] Wang J, Zhang K, Liu T, Song Y, Hua P, Chen S, Li J, Liu Y, Zhao Y. Efficacy and safety of neoadjuvant immunotherapy combined with chemotherapy in locally advanced esophageal cancer: A meta-analysis. Front Oncol. 2022 Sep 5;12:974684. doi: 10.3389/fonc.2022.974684. eCollection 2022. PMID 36158679
- [Result] Yang Y, Liu J, Liu Z, Zhu L, Chen H, Yu B, Zhang R, Shao J, Zhang M, Li C, Li Z. Two-year outcomes of clinical N2-3 esophageal squamous cell carcinoma after neoadjuvant chemotherapy and immunotherapy from the phase 2 NICE study. J Thorac Cardiovasc Surg. 2024 Mar;167(3):838-847.e1. doi: 10.1016/j.jtcvs.2023.08.056. Epub 2023 Sep 9. PMID 37696429
- [Result] Yan X, Duan H, Ni Y, Zhou Y, Wang X, Qi H, Gong L, Liu H, Tian F, Lu Q, Sun J, Yang E, Zhong D, Wang T, Huang L, Wang J, Chaoyang Wang, Wang Y, Wan Z, Lei J, Zhao J, Jiang T. Tislelizumab combined with chemotherapy as neoadjuvant therapy for surgically resectable esophageal cancer: A prospective, single-arm, phase II study (TD-NICE). Int J Surg. 2022 Jul;103:106680. doi: 10.1016/j.ijsu.2022.106680. Epub 2022 May 18. PMID 35595021

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT06364566/SAP_000.pdf